CLINICAL TRIAL: NCT06301815
Title: Identifying Vertical Perception Loss in People With Acute Stroke: A Feasibility Study
Brief Title: Feasibility of Measuring Vertical Perception in Acute Stroke
Status: Completed | Type: Observational
Sponsor: University of Winchester (Other)
Collaborators: Hampshire Hospitals NHS Foundation Trust (Other); University Hospitals Dorset NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: Shaw_Stroke_REC24/YH/0010_2024
Record Dates: First submitted 2024-03-03; First posted 2024-03-08 (Actual); Results first posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Stroke
Keywords: Vertical Perception; Rehabilitation; Neglect; Pushing Behaviour; Subjective Visual Vertical
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Scale for Contraversive Pushing — Lateropulsion will be assessed using the Scale for Contraversive Pushing (SCP). It involves observation of the posture of the participant in sitting and standing. Scores are assessed in sitting and standing giving a maximum score of 6.
Diagnostic Test: Catherine Bergego Scale — Neglect will be assessed using the Catherine Bergego Scale. The scale is a 10-point scale with each item scored between 0 (no neglect) and 3 (severe neglect). It involves observation of a participant completing daily activities such as eating, dressing and walking.
Diagnostic Test: Bucket Test — The bucket test involves the patient being sat upright and looking into a translucent bucket with the bucket covering their complete field of vision. On the inside of the bucket on the bottom is a dark straight line. On the outside of the bottom of the bucket is a matching dark line, the bottom of the bucket is divided into degrees with the zero-degree line being equivalent to the line inside the bucket. For measurement the bucket will be randomly rotated right or left by the examiner to 45 degrees and then slowly rotated back to the zero-degree position. Patients will signal when they estimate the inside bottom line to be truly vertical by saying "stop" or by raising their non-paretic hand.

SUMMARY:
The goal of this observational study is to establish if it is feasible to identify vertical perception deficits in people with acute stroke. The primary purpose to the study is:

• To establish the feasibility of completing the Catherine Bergego Scale, Scale for Contraversive Pushing (SCP) and bucket test in a clinical environment with acute stroke patients to assist with identification of vertical perception loss.

Participants will be asked to complete the assessments with a therapist 48 hours after admission. If they are not completed for any reason attempts will be made to complete them at one, two and four weeks after admission. Some participants will have them completed again on discharge. The Catherine Bergego Scale and SCP are observational and will involve a therapist watching the participant undertake daily activities. The bucket test involves a therapist placing a bucket in front of the face of the participant and asking them to identify when a line on the bottom of the bucket is vertical. Acceptabiliy and feasibility will be further investigated using a survey of participants who complete the assessments and through focus groups with the rehabilitation professionals admininstering the assessments.

If it is feasible and acceptable to complete these assessments then further research can use them as an acceptable measure of vertical alignment in the clinical setting.

DETAILED DESCRIPTION:
The secondary research questions that this study will aim to address are:

* What percentage of patients admitted to an acute stroke unit show a positive test for vertical perception loss within four weeks of admission (evidence of subjective visual vertical (SVV) tilt on either bucket test or Catherine Bergego Scale or evidence of subjective postural vertical (SPV) tilt on SCP)?
* For those able to complete the assessments, does vertical perception loss show any relationship with:

  * Discharge (DC) destination
  * Care package size on discharge
  * Number of inpatient falls
  * Level of functional independence on discharge
* Is there a trend for any element of the SCP or the Catherine Bergego to be more correlated with SVV tilt.

Primary outcomes:

The primary outcome is to understand the feasibility of completing the suite of outcome measures in an acute stroke setting. The study will determine the :

* Proportion (%) of patients on whom the assessments are attempted.
* Percentage of patients who are able to complete all three assessments within four weeks of admission.
* Time taken to complete the three measures in an acute clinical setting
* A recommendation regarding the most feasible time point to complete these assessments.

Secondary outputs:

The secondary aims are to gain a further understanding of vertical perception loss in acute stroke patients.

* An understanding of factors that prevent or facilitate completion of these three assessments
* An understanding of healthcare professionals' experiences of completing these assessments in an acute stroke unit.
* An understanding of whether people with stroke (or their advocates) find it appropriate to complete all three assessments in an acute stroke setting.
* Percentage of patients admitted to an acute stroke unit showing a positive test for vertical perception loss within four weeks of admission.
* To explore the relationship between vertical perception loss and:

  * Discharge destination
  * Care package size on discharge
  * Number of inpatient falls
  * Level of functional independence on discharge
* To explore if any elements of the Catherine Bergego Scale or Scale for Contraversive Pushing show a trend for a relationship to vertical perception loss Trial Setting The population to be studied will be acute stroke patients admitted to a stroke unit. A non-probability, convenience sample will be used. All patients with a diagnosis of stroke admitted for 72 hours to a single stroke unit at Royal Hampshire County Hospital will be considered in the present study. All those admitted to the stroke unit over a six-month period will be eligible for inclusion, meaning approximately 250 people will be screened for participation.

Recruitment Potential participants will be identified during the daily handover. Those meeting the inclusion criteria will be approached and invited to participate. This will take place between 48 hours and one week after admission. Potential participants will be provided with the participant information sheet (PIS). If the patient is unable to consent due to cognitive or language impairment or low level of consciousness then their advocate will be approached. Where possible potential participants will be supported to consent using information in different formats (e.g. through use of pictures) or the skill of appropriate members of the clinical team (e.g. speech and language therapists).

If a participant who lacked capacity, and was consented by an advocate, regains capacity then their informed consent to continue will be sought.

Study protocol For those patients who consent, the qualified physiotherapists or occupational therapists on the stroke unit, will then attempt to complete all 3 outcome measures with the patient. If the patient is unable to complete any elements of the outcome measure for any reason, this will be recorded. If the patient is unable to complete the outcome measures, then an attempt will be made to complete the outcome measures at 1 week post admission, if still unable they will be attempted again at 2 weeks and 4 weeks post admission. At the point participants complete all 3 outcome measures or at 4 weeks (whichever is earliest) most will have no further active participation in the quantitative part of the study. The assessments do not need to all be completed in one sitting and can be spread across sessions. If a patient is unable to be consented at 48 hours they will be consented as soon after this point as possible up to one week after admission, and this will be recorded. If patients are discharged or have a change in status following consenting to participate but prior to completion of the outcome measures any data collected to date will be utilised in the study results and the reasons for non-completion of the outcome measures will be noted as this will inform the feasibility of these outcome measures. The length of time taken to complete the measures will be recorded by the administrator. The expectation is that administration of all three outcome measures will take no longer than one hour. Due to the observational nature of the SCP and Catherine Bergego Scale elements of these can be completed during therapy sessions.

At the point the participants are discharged from the stroke unit appropriate information will be extracted from their medical records.

At the time of discharge a small sub-selection of the study participants will have the outcome measures reassessed. Participants will be identified as having a mild, moderate or severe vertical perception loss in order to allow a spectrum of loss to be measured during inpatient stay. Once discharged from the stroke unit participants will have no further input into the study.

Assessors Outcome measures will be undertaken by a qualified member of the therapy team on the stroke unit. This includes physiotherapists and occupational therapists. All those undertaking the outcome measures will be trained on their use by the main author (AS) to ensure consistency of approach.

Additional Research Activities. Focus Groups Prior to the study commencing a focus group will be completed with the therapists undertaking the outcome measures. This will be held following training on the outcome measures. Therapists will be invited to attend by AS at the end of the training session and provided with a PIS.

This will allow exploration of how feasible or acceptable the therapists feel it will be to complete the outcome measures before data collection. This can then be compared with their thoughts, and the thoughts of people with stroke and their advocates, on acceptability following use of the outcome measures.

At the six month point of the study the focus group will be repeated, with approximately 10 therapists, to allow exploration of the experiences of the therapists that undertook the outcome measures. This will allow collection of data from multiple participants using an unstructured but guided discussion of the use of the outcome measures in the acute stroke setting.

Potential participants will be members of the therapy team on the stroke unit who have undertaken the outcome measures.They will be provided with a PIS explaining the post-trial focus groups and the time and date at which the group will be undertaken. They can then decide if they wish to participate or not.

If they wish to participate they will be asked to sign a consent form and attend the group at the dedicated time. The groups will be moderated by the lead researcher (AS) using a list of topics/questions to guide the conversation. A second member of the research team, unknown to the participants, will assist in the groups to ensure smooth running of the groups and mitigate for the fact that AS will be known to many participants. Face to face groups will be held in the hospital setting at a time convenient to a majority of participants. The focus groups will last no longer than 1.5 hours. Ground rules will be introduced at the beginning of the groups to allow smooth running of the group and to put participants at ease. Focus groups will be recorded for transcription on MS Teams and stored behind two factor authentication on a password protected computer. Each group member will be assigned a participant number to assist with data analysis. The focus group will be anonymised and transcribed verbatim and following transcription the original recording will be deleted. At this point participants will no longer be able to withdraw from the study.

Patient Participant Feedback At the point they complete all the outcome measures (or at 4 weeks if they are unable to complete the measures) participants (or their advocates) will be asked to complete a short survey asking about the acceptability of the outcome measures. Questions will ask about their attitude towards, understanding of and burden of completing the outcome measures. It will be a mix of choice and Likert scale questions with some free text open questions. The survey should take no more than 15 mins to complete. Participants can be supported to complete the survey by an advocate, therapist or member of the research team who can read out the questions and record their responses, but will not influence the answers. The survey will be on paper for ease of completion in the clinical setting.

The decision as to whether it is feasible to use these outcome measures to identify those with vertical perception loss will be made on the basis of collated results of this trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of first stroke by stroke consultant based on clinical or radiographical findings
* Admitted to stroke unit with a length of stay of over 72 hours
* Ability to consent or an advocate to consent on their behalf
* Pre-morbid Modified Rankin Scale of less than 4

Exclusion Criteria:

* Under the age of 18
* Diagnosis of Transient Ischaemic Attack (TIA)
* Previous diagnosis of stroke or other neurological diagnosis affecting the brain with residual impairment
* Patients on an end of life pathway
* Patients with pre-morbid visual impairment that will not allow them to see the bucket test. Glasses can be worn.
* Inability to speak the English language and no interpreter can be found

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute stroke patients in inpatient care
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof James Faulkner, PhD, Study Director — University of Winchester
Locations (1):
- Royal Hampshire County Hospital, Winchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between 1/5/2024 and 31/10/2024 on the acute stroke unit at Hampshire Hospitals NHS Foundation Trust, UK.
Pre-assignment Details: No significant Events
Groups:
- Intervention Group: Participants who underwent the interventions as laid out in the protocol. As this was an observational study all participants underwent three assessments (bucket test, Catherine Bergego Scale and Scale for contraversive pushing) once on recruitment. There was only one group. These assessments were completed as soon as possible after admission to an acute stroke unit and were all completed by four weeks.
Period: Overall Study
Arm/Group | Intervention Group
Started | 53 (01/05/2024)
Completed | 53 (30/10/2024)
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Intervention Group: Participants who underwent the interventions as laid out in the protocol
Arm/Group | Intervention Group
Number analyzed (Participants) | 53
Age, Continuous [Mean (Full Range); unit: Years] | 77 [45 to 99]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Bucket Test to Measure Subjective Visual Vertical (SVV).
Description: The bucket test involves the patient being sat upright and looking into a translucent bucket. On the inside of the bucket on the bottom is a dark straight line. On the outside of the bottom of the bucket is a matching dark line, the bottom of the bucket is divided into degrees with the zero-degree line being equivalent to the line inside the bucket. For measurement the bucket will be randomly rotated right or left by the examiner to 45 degrees and then slowly rotated back to the zero-degree position. Patients will signal when they estimate the inside bottom line to be truly vertical by saying "stop" or by raising their non-paretic hand. Degrees will be read off on the outside scale by the examiner. The procedure will be repeated 6 times (3 to left and 3 to right) in a random order. A mean of the 6 tests will be calculated to be the tilt of SVV. The standard deviation (SD) of the mean of the 6 tests will be calculated to represent the uncertainty of SVV.
Time Frame: Admission, 1 week, 2 weeks and 4 weeks, but not repeated once successfully completed.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Intervention Group
Number analyzed (Participants) | 53
Degrees | 3.2 (3.6)

2. Primary Outcome: Catherine Bergego Scale to Measure Neglect.
Description: Neglect will be assessed using the Catherine Bergego Scale. This established outcome measure for neglect is free and observational, it reflects existing practice and therefore reduces the burden on research participants. The scale is a 10-point scale with each item scored between 0 (no neglect) and 3 (severe neglect). Such as grooming, walking, eating and dressing. Minimum score is 0 - no neglect and maximum score is 30 - severe neglect
Time Frame: Admission, 1 week, 2 weeks and 4 weeks, but not repeated once successfully completed.
Measure: Median (Inter-Quartile Range); unit: Units on a scale (0-30)
Arm/Group | Intervention Group
Number analyzed (Participants) | 53
Units on a scale (0-30) | 0 [0 to 1]

3. Primary Outcome: Scale for Contraversive Pushing to Measure Lateropulsion
Description: Lateropulsion will be assessed using the Scale for Contraversive Pushing (SCP). This observational assessment can be conducted as part of routine therapy sessions. Scores are assessed in sitting and standing giving a maximum score of 6. The SCP has been found to be a reliable and valid measure. It involves observation of the posture of the patient in sitting and standing. Minimum score of 0 is no sign of lateropulsion and maximum score of 6 is severe lateropulsion.
Time Frame: Admission, 1 week, 2 weeks and 4 weeks, but not repeated once succesfully completed.
Measure: Median (Inter-Quartile Range); unit: Units on a scale (0-6)
Arm/Group | Intervention Group
Number analyzed (Participants) | 53
Units on a scale (0-6) | 0 [0 to 1]

ADVERSE EVENTS:
Time Frame: From enrollement until study end - 4 weeks
Description: As per the clinicaltrials.gov definitions
Arm/Group | Intervention Group
All-Cause Mortality (participants affected / at risk) | 1/53
Serious Adverse Events (participants affected / at risk) | 0/53
Other Adverse Events (participants affected / at risk) | 0/53

LIMITATIONS AND CAVEATS:
No known limitations or caveats

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-09): https://cdn.clinicaltrials.gov/large-docs/15/NCT06301815/Prot_SAP_000.pdf
  • Informed Consent Form (2024-01-24): https://cdn.clinicaltrials.gov/large-docs/15/NCT06301815/ICF_001.pdf